CLINICAL TRIAL: NCT06675955
Title: An Open-Label, Multicenter Extension Study Evaluating the Patient Perspective of the Physical Impact of Multiple Sclerosis and Providing Continued Access to Ocrelizumab in Patients With Multiple Sclerosis Previously Enrolled in a Genentech and/or F. Hoffmann-La Roche Ltd Sponsored Study and Without Access to a Post-Trial Access Program
Brief Title: An Extension Study to Assess Impact of Multiple Sclerosis (MS) on Physical Function and Provide Continued Ocrelizumab Treatment
Acronym: OleroMAX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MN45053; 2023-507633-21-01 (EU CTIS Number)
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
Keywords: Ocrelizumab
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ocrelizumab (Experimental): Participants will receive ocrelizumab at the same dose and schedule as the parent study until access to the treatment becomes locally available, unacceptable safety concern, death or withdrawal of consent.
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Ocrelizumab will be administered according to the regimen in the parent study.
  Other Names: RO4964913

SUMMARY:
The study will evaluate the physical impact of MS from participant's perspective, provide continued access to ocrelizumab and assess the safety and tolerability of ocrelizumab.

ELIGIBILITY:
Inclusion Criteria:

* Participants who were on ongoing ocrelizumab treatment on one of the following parent-studies [Studies MN39159/CONSONANCE (NCT03523858), BN42082/MUSETTE (NCT04544436), BN42083/GAVOTTE (NCT04548999), BN44083/GLOBEAM, MN43978/CONSONANCE Ext., WA40404/O'HAND (NCT04035005), MN43964/OLERO (NCT05269004), GN41791/FENTREPID (NCT04544449), BP46016/MINTAKA, CN41144/OCARINA I-SC (NCT03972306), CN42097/OCARINA II-SC (NCT05232825)] at the time of roll-over and who do not have access to the ocrelizumab treatment locally.
* The first dose of study treatment in this extension study will be received no earlier than 5 months after the last treatment in the parent study.
* Negative urine pregnancy test within 24 hours to first dose administered on MN45053 study treatment in participants of childbearing potential.

Exclusion Criteria:

* Study treatment is commercially marketed in the participant's country for the participant specific disease and is reasonably accessible to the participant.
* Study treatment is available via Post Trial Access Program (PTAP) in the participant's country and is accessible to the participant.
* Permanent premature discontinuation of study treatment for any reason during the parent study or during the time between last treatment in the parent study and the first dose of study treatment in this extension study (if applicable).
* Any condition that, in the opinion of the investigator, would interfere with the interpretation of participant safety or place the participant at high risk for treatment-related complications.
* Concurrent participation in any therapeutic clinical trial (other than the parent study).
* Immunocompromised state
* Known active malignancy or are being actively monitored for recurrence of malignancy.
* Known presence of other neurological disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline to End of Study in the Physical Functioning Score of the Patient-Reported Outcome Measure Information System/Quality of Life in Neurological Disorders-Physical Function Measure for Multiple Sclerosis 15a (PROMISnq PFMS-15a) | Baseline up to 5 years
  PROMISnq PFMS-15a includes 15 items that evaluate the impact of MS on a participant's physical functioning, including mobility, upper limb function and activities of daily living. Nine items assess the degree of difficulty in completing physical activities using a 5 point verbal rating scale ranging from 5="without any difficulty" to 1="unable to do". Four items assess physical function limitations, rated from 5="not at all" to 1="cannot do". Two items assess the amount of difficulty associated with selected physical activities, rated from 5="no difficulty" to 1="can't do". Scores are reported as a standardized T-score metric, with higher scores reflecting better physical functioning.
Number of Eligible Participants who Have Received Access to Ocrelizumab in the Study | Up to 5 years

SECONDARY OUTCOMES:
Number of Participants with Serious Adverse Events (SAEs) | Up to 5 years
Number of Participants with Adverse Events (AEs) Leading to Discontinuation | Up to 5 years
Number of Participants with Adverse Events of Special Interest (AESIs) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (41):
- France (12):
  - CHU Amiens Hopital Sud, Amiens Cedex1
  - CHU de Besancon Hopital Jean Minjoz, Besançon
  - Groupe Hospitalier Pellegrin, Bordeaux
  - CHU Brest Hopital La Cavale Blanche, Brest
  - Hopital neurologique Pierre Wertheimer - CHU Lyon, Bron
  - CHU De Caen, Caen
  - Hopital Gabriel Montpied CHU de Clermont-Ferrand, Clermont-Ferrand
  - CH St Vincent de Paul, Lille
  - Hopital Gui de Chauliac, Montpellier
  - Hôpital Pasteur, Nice
  - GroupeHospitalo-Universitaire Caremeau, Nîmes
  - Hopital de Hautepierre, Strasbourg
- Germany (3):
  - NeuroPoint Gesellschaft fur vorbeugende Gesundheitspflege mbH, Ulm
  - Studienzentrum Nordwest Dr med Joachim Springub Herr Wolfgang Schwarz, Westerstede
  - Deutsche Klinik für Diagnostik, Wiesbaden
- Russia (14):
  - Krasnoyarsk State Medical Academy, Krasnoyarsk, Krasnoyarsk Krai
  - FSBHI Siberian Clinical Center of the Federal Medical and Biological Agency, Krasnoyarsk, Krasnoyarsk Krai
  - City Clinical Hospital #24, Moscow, Moscow Oblast
  - Federal center of brain research and neurotechnologies, Moskva, Moscow Oblast
  - LLC Osnova, Saint Petersburg, Sankt-Peterburg
  - N.P. Bechtereva Institute of the Human Brain, Saint Petersburg, Sankt-Peterburg
  - City Hospital #40 of Kurortniy Administrative District, Saint Petersburg, Sankt-Peterburg
  - SHI Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg, Sverdlovsk Oblast
  - Vertebronevrologiya LLC, Kazan', Tatarstan Republic
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk, Ulyanovsk Oblast
  - Center of Cardiology and Neurology, Kirov
  - Regional clinical hospital named after prof. S.V. Ochapovsky, Krasnodar
  - FSBIH Siberian Regional Medical Centre of FMBA of Russia, Novosibirsk
  - Perm SMA n.a. academ. E.A. Vagner, Perm
- Ukraine (12):
  - 5th Cherkasy City Center of Primary Health Care, Cherkasy
  - Mun.Med.Proph.Inst.?Chernihiv Reg.Hosp.?, Chernihiv
  - Bukovinsky SMU RMI Chernivtsi RCH, Chernivtsi
  - SI USSRI of Medical and Social Problems of Disabilities of MOHU, Dnipro
  - Regional Clinical Hospital, Ivano-Frankivsk
  - St.In.Inst. of Neurol.Psych.and Narcol.of the AMSU, Kharkiv
  - Medical Center Dopomoga Plus, Kyiv
  - Medical Center of Private Execution First Private Clinic, Kyiv
  - Lvivska oblasna tsentralna likarnia, Lviv
  - Medical Clinical Research Center of Medical Center LLC Health Clinic, Vinnytsi
  - LCC "Medical center "Unimed", Zaporizhzhia
  - Municipal Non-profit Enterprise Zaporizhzhya Regional Hospital Zaporizhzhya Regional Council, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing